CLINICAL TRIAL: NCT05458232
Title: Use of a Phosphodiesterase Type 5 Inhibitor to Improve Anabolic Resistance in Older Adults
Status: Withdrawn | Type: Observational
Why Stopped: No subjects enrolled
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 273780
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2022-12

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Tadalafil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood/plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 5mg tadalafil once daily for 14 days
  Interventions: Drug: Tadalafil 5mg

INTERVENTIONS:
Drug: Tadalafil 5mg — Subjects will ingest one 5mg tablet of tadalafil each evening for 14 days.

SUMMARY:
This study will be the first demonstration of the utility and feasibility of Phosphodiesterase Type 5 inhibitor as an effective pharmacological therapy for improving anabolic resistant states.

ELIGIBILITY:
Inclusion Criteria:

* Ages 60-75 yrs
* Recently prescribed 5mg of tadalafil daily for clinical purposes

Exclusion Criteria:

* History of diabetes
* history of hypotension including orthostatic hypotension
* History of malignancy or chemo/radiation therapy in the 6 months prior to enrollment
* History of short gut syndrome, gastrointestinal bypass/reduction surgery (Lap band, gastric sleeve, etc.)
* Subjects who cannot refrain from using protein or amino acid supplements for 7 days prior to Visit 2 and 3.
* Alcohol consumption of ≥ 5 units/servings per day
* Concomitant use of

  * oral or injectable corticosteroids
  * testosterone, insulin like growth factor-1, or similar anabolic agent
  * riociguat (Adempas)
  * nitroglycerin
  * isosorbide dinitrate (Isordil)
  * isosorbide mononitrate (Imdur, Monoket)
  * doxazosin (Cardura)
  * prazosin (Minipress)
  * terazosin (Hytrin)
* Any other disease or condition that would place the subject at increased risk of harm if they were to participate, at the discretion of the study physician

Ages: 60 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males 60-75 years who have been prescribed 5mg daily tadalafil by their physician.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Change in maximal voluntary contraction of lower leg. | 14 days
  Lower leg strength using a dynamometer; performed both before and after 14 days of tadalafil

SECONDARY OUTCOMES:
Change in muscle Fatigue | 14 days
  A test of lower leg muscular endurance using a dynamometer; performed both before and after 14 consecutive days of tadalafil.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenberg IH. Sarcopenia: origins and clinical relevance. J Nutr. 1997 May;127(5 Suppl):990S-991S. doi: 10.1093/jn/127.5.990S. PMID 9164280